CLINICAL TRIAL: NCT06802198
Title: Comparison of Long-Term Outcomes Following Laparoscopic Total Vs Supracervical Hysterectomy, a Randomized Clinical Trial
Brief Title: A Randomized Study Comparing Subtotal vs Total Hysterectomy Long Term Outcomes
Acronym: STORY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6429
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-01

CONDITIONS: Fibroid Uterus; Metrorrhagia; Adenomyosis; Benign Gynecologic Neoplasm; Endometriosis; Abnormal Uterine Bleeding
MeSH Terms: conditions — Leiomyoma; Metrorrhagia; Adenomyosis; Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients undergoing total hysterectomy (Active Comparator): Total hysterectomy involves the complete removal of the uterus including the cervix
  Interventions: Procedure: total hysterectomy
- patients undergoing subtotal hysterectomy (Experimental): Subtotal hysterectomy involves the removal of the upper part of the uterus preserving the cervix
  Interventions: Procedure: subtotal hysterectomy

INTERVENTIONS:
Procedure: total hysterectomy — Total hysterectomy (TH) involves the complete removal of the uterus including the cervix
  Arms: patients undergoing total hysterectomy
Procedure: subtotal hysterectomy — subtotal hysterectomy (STH) preserves the cervix while removing the upper part of the uterus
  Arms: patients undergoing subtotal hysterectomy

SUMMARY:
The goal of this randomized clinical trial is to assess the outcomes of total laparoscopic hysterectomy vs subtotal laparoscopic hysterectomy + mini-laparotomy for uterine extraction for benign gynecological conditions in terms of change in quality of life at 36 months after surgery and patient's impression of improvement. The secondary objectives of the study are to assess any differences in terms of peri and postoperative outcomes (postoperative pain, blood loss, hospital stay, intraoperative or short and long-term postoperative complications, long term urinary, bowel and pelvic floor symptoms, prevalence of vaginal cuff dehiscence).

Participants will fill the following questionnaires pre-operatively and at the follow up:

* Short Form 36 (SF36),
* Euro Quality of life 5D-3L (EQ 5D-3L)
* Female Sexual Function Index (FSFI)
* Patient Global Impression of Improvement (PGI-I) only during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Signed informed consent

Exclusion Criteria:

* Uterine or adnexal pathology suspect for malignancy
* Abnormal or unknown PAP test
* Patients with invasive neoplasia in the previous 5 years (excluding non-melanoma skin tumors, breast cancer T1 N0 M0 Grade 1 or 2 without signs of recurrence or activity).
* Previous radical pelvic surgery or radiotherapy;
* Age > 80 years
* Pregnant patients
* Desire for further pregnancies
* Contraindications to general anaesthesia or to the Trendelenburg position
* Refusal to sign informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life and patient's impression of improvement at 36 months after surgery | 5 years
  To assess the impact of surgery on patients' quality of life measured by the Physical Functioning items of SF36 questionnaire, at 36 months after surgery

SECONDARY OUTCOMES:
Postoperative pain | 5 years
  Post-operative pain will be evaluated using the visual analog scale (VAS) score, every 6 hours from the end of surgery, up to 48 hours.
Intra-operative data | 5 years
  To compare of operative time, estimated blood loss, associated procedures, and need for conversion to other techniques.
intraoperative complications | 5 years
  To evaluate the occurrence of intraoperative complications according to the modified Satava classification system. Grade 1 complications include incidents without consequences for the patient; grade 2 complications, which are treated intraoperatively with endoscopic surgery (grade 2a) or required endoscopic re-treatment (grade 2b); and grade 3 complications include incidents requiring open or laparoscopic surgery.
short and long-term postoperative complications | 5 years
  To evaluate the occurrence of postoperative complications according to the Clavien-Dindo classification and to evaluate the occurrence of long-term complications, including vaginal cuff dehiscence, up to 36 months post-operatively
Urinary, bowel and pelvic floor symptoms | 5 years
  To evaluate the impact of surgery on other urinary and bowel symptoms, with particular attention to 'de novo' symptoms, and long-term occurrence of pelvic organ prolapse or pelvic floor dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Panico, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Ginecologia Oncologica, Rome, Lazio, Italy